CLINICAL TRIAL: NCT06586684
Title: The Effect of Small Interfering RNA Inclisiran on Carotid Plaques in Patients with Atherosclerosis: a Real-world Study Using Carotid Ultrasound.
Brief Title: Effect of Small Interfering RNA Inclisiran on Carotid Plaques As Assessed by Carotid Ultrasound
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Zhenyan Fu, PHD, Pricinple Inverstigator, First Affiliated Hospital of Xinjiang Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EICP-UCG
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Carotid Plaque; Hyperlipidemia; Echocardiography
Keywords: inclisiran; carotid plaque; Echocardiography; hyperlipidmia
MeSH Terms: conditions — Hyperlipidemias | interventions — ALN-PCS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- inclisiran Therapy group (Experimental): Patients with carotid plaques undergoing treatment with inclisiran
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Drug: Inclisiran — Patients with carotid plaques undergoing treatment with inclisiran

SUMMARY:
Current understanding suggests that the majority of cardiovascular events are driven by vulnerable plaques. Nonetheless, the impact of PCSK9 inhibitors on the stability of carotid plaques remains insufficiently elucidated, with a notable scarcity of relevant clinical studies. This investigation seeks to address this gap through a real-world study conducted among patients with arterial sclerosis in Asia. The primary aim is to evaluate the effects of small interfering RNA (inclisiran) on carotid plaque characteristics as assessed by ultrasound, thereby contributing valuable data to inform clinical practice.

DETAILED DESCRIPTION:
In a meticulous study evaluating the impact of inclisiran on patients with atherosclerosis and carotid plaques, data were systematically gathered across multiple time points. The assessment encompassed:Blood Samples: Analyzed at baseline (Month 0) and subsequently at Months 1, 2, 3, 5, 9, 11, and 12, examining biochemical markers, lipid profiles, and liver and kidney function tests.Carotid Ultrasound: Conducted at Months 0, 3, 9, and 12, monitoring the carotid intima-media thickness, maximum carotid plaque thickness, carotid plaque area, carotid plaque volume, and carotid lumen stenosis area for thorough analysis.Clinical Records: Documented in detail the baseline clinical information, biochemical markers, imaging findings, and any adverse cardiovascular or cerebrovascular events that occurred throughout the study period. This approach ensures a comprehensive understanding of inclisiran's effects over time, encompassing both biochemical and imaging parameters, while tracking potential adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid plaques as indicated by ultrasound
* Men and women aged 18-75 years;
* LDL-C >3.4 mmol/L without regular statin therapy or LDL-C >1.8 mmol/L after 4 weeks of statin lipid-lowering therapy.

Exclusion Criteria:

* - Known allergies or contraindications to PCSK9 inhibitors and/or statin therapy;
* Prior use of PCSK9 inhibitors;
* Prior history of hemorrhagic stroke;
* Prior coronary artery bypass grafting or coronary intervention;
* Inability to perform OCT imaging or unclear imaging;
* Severe renal insufficiency (creatinine clearance < 30 mL/min);
* Severe hepatic dysfunction;
* Baseline triglycerides > 5.6 mmol/L;
* Pregnant or lactating women;
* Life expectancy not exceeding 1 year;
* In the judgment of the investigator, unsuitable for this study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
CIMT | Immediately and treated with inclisiran one year later
  Carotid artery intima media thickness
TMPT | Immediately and treated with inclisiran one year later
  The maximal plaque thickness
CPA | Immediately and treated with inclisiran one year later
  Carotid plaque area
CPV | Immediately and treated with inclisiran one year later
  Carotid plaque volume
CALA | Immediately and treated with inclisiran one year later
  Carotid artery lumen area

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyan Fu, PhD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University

IPD SHARING:
Plan to Share IPD: No
IPD will be made available on reasonable request to the official agencies.

REFERENCES:
- [Background] Ray KK, Wright RS, Kallend D, Koenig W, Leiter LA, Raal FJ, Bisch JA, Richardson T, Jaros M, Wijngaard PLJ, Kastelein JJP; ORION-10 and ORION-11 Investigators. Two Phase 3 Trials of Inclisiran in Patients with Elevated LDL Cholesterol. N Engl J Med. 2020 Apr 16;382(16):1507-1519. doi: 10.1056/NEJMoa1912387. Epub 2020 Mar 18. PMID 32187462
- [Background] Wright RS, Ray KK, Raal FJ, Kallend DG, Jaros M, Koenig W, Leiter LA, Landmesser U, Schwartz GG, Friedman A, Wijngaard PLJ, Garcia Conde L, Kastelein JJP; ORION Phase III Investigators. Pooled Patient-Level Analysis of Inclisiran Trials in Patients With Familial Hypercholesterolemia or Atherosclerosis. J Am Coll Cardiol. 2021 Mar 9;77(9):1182-1193. doi: 10.1016/j.jacc.2020.12.058. PMID 33663735
- [Background] Huo Y, Lesogor A, Lee CW, Chiang CE, Mena-Madrazo J, Poh KK, Jeong MH, Maheux P, Zhang M, Wei S, Han Y, Li Y. Efficacy and Safety of Inclisiran in Asian Patients: Results From ORION-18. JACC Asia. 2023 Nov 14;4(2):123-134. doi: 10.1016/j.jacasi.2023.09.006. eCollection 2024 Feb. PMID 38371290
- [Background] Mantella LE, Colledanchise KN, Hetu MF, Feinstein SB, Abunassar J, Johri AM. Carotid intraplaque neovascularization predicts coronary artery disease and cardiovascular events. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1239-1247. doi: 10.1093/ehjci/jez070. PMID 31621834
- [Background] Wong EY, Nikolov HN, Rankin RN, Holdsworth DW, Poepping TL. Evaluation of distal turbulence intensity for the detection of both plaque ulceration and stenosis grade in the carotid bifurcation using clinical Doppler ultrasound. Eur Radiol. 2013 Jun;23(6):1720-8. doi: 10.1007/s00330-012-2741-6. Epub 2012 Dec 18. PMID 23247808
- [Background] Wright RS, Collins MG, Stoekenbroek RM, Robson R, Wijngaard PLJ, Landmesser U, Leiter LA, Kastelein JJP, Ray KK, Kallend D. Effects of Renal Impairment on the Pharmacokinetics, Efficacy, and Safety of Inclisiran: An Analysis of the ORION-7 and ORION-1 Studies. Mayo Clin Proc. 2020 Jan;95(1):77-89. doi: 10.1016/j.mayocp.2019.08.021. Epub 2019 Oct 17. PMID 31630870
- [Background] Crouse JR 3rd, Raichlen JS, Riley WA, Evans GW, Palmer MK, O'Leary DH, Grobbee DE, Bots ML; METEOR Study Group. Effect of rosuvastatin on progression of carotid intima-media thickness in low-risk individuals with subclinical atherosclerosis: the METEOR Trial. JAMA. 2007 Mar 28;297(12):1344-53. doi: 10.1001/jama.297.12.1344. Epub 2007 Mar 25. PMID 17384434
- [Background] Wu L, Kong Q, Huang H, Xu S, Qu W, Zhang P, Yu Z, Luo X. Effect of PCSK9 inhibition in combination with statin therapy on intracranial atherosclerotic stenosis: A high-resolution MRI study. Front Aging Neurosci. 2023 Mar 9;15:1127534. doi: 10.3389/fnagi.2023.1127534. eCollection 2023. PMID 36967822
- [Background] Ray KK, Kallend D, Leiter LA, Raal FJ, Koenig W, Jaros MJ, Schwartz GG, Landmesser U, Garcia Conde L, Wright RS; ORION-11 Investigators. Effect of inclisiran on lipids in primary prevention: the ORION-11 trial. Eur Heart J. 2022 Dec 21;43(48):5047-5057. doi: 10.1093/eurheartj/ehac615. PMID 36331315
- [Background] Chen J, Zhao F, Lei C, Qi T, Xue X, Meng Y, Zhang W, Zhang H, Wang J, Zhu H, Cheng C, Wang Q, Bi C, Song B, Jin C, Niu Q, An F, Li B, Huo X, Zhao Y, Li B. Effect of evolocumab on the progression of intraplaque neovascularization of the carotid based on contrast-enhanced ultrasonography (EPIC study): A prospective single-arm, open-label study. Front Pharmacol. 2023 Jan 4;13:999224. doi: 10.3389/fphar.2022.999224. eCollection 2022. PMID 36686711
- [Background] Aranzulla TC, Piazza S, Ricotti A, Musumeci G, Gaggiano A. CARotid plaqUe StabilizatiOn and regression with evolocumab: Rationale and design of the CARUSO study. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):E115-E121. doi: 10.1002/ccd.29743. Epub 2021 Apr 24. PMID 33893754